CLINICAL TRIAL: NCT03463824
Title: The VIGOR Study - Virtual Immersive Gaming to Optimize Recovery in Low Back Pain
Acronym: VIGOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Ohio University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20014058; 1R01HD088417-01A1 (NIH); 17-F-11 (Other: Ohio University)
Record Dates: First submitted 2018-02-13; First posted 2018-03-13 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low Back Pain; Fear of Pain; Fear of Injury

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two intervention arms. Both intervention arms involve immersive video games that encourage participants to produce progressively larger lumbar flexion excursions at each game level and across treatment sessions. The two groups are distinguished by the amount of lumbar flexion needed to achieve game objectives. One is a control group and the other is the experimental.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The principal investigators, the statistician, and members of the data collection team will remain blinded to intervention assignment throughout the duration of the study. They will be given the identifying codes only at the end of the study when it is necessary to interpret the results. The un-blinded study coordinator, who is responsible for scheduling testing and treatment sessions, will serve to receive the study patients and escort them to the various testing and treatments sites to minimize the interaction between patients; however, the study coordinator will not participate in the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants will produce progressively larger lumbar flexion excursions at each game level and across treatment sessions. The control group will play the same immersive video games, but the parameters will be modified such that only small excursions of lumbar flexion are needed to successfully complete gameplay.
  Interventions: Behavioral: Experimental Group 1
- Experimental Group 2 (Experimental): Participants will produce progressively larger lumbar flexion excursions at each game level and across treatment sessions.
  Interventions: Behavioral: Experimental Group 2

INTERVENTIONS:
Behavioral: Experimental Group 1 — Participants will complete 18 intervention visits over 9 weeks with the number of sessions tapered across weeks (i.e., 3 sessions/week in weeks 1-3, 2 sessions/week in weeks 4-6, and 1 session/week in weeks 7-9).
  Arms: Control Group
Behavioral: Experimental Group 2 — Participants will complete 18 intervention visits over 9 weeks with the number of sessions tapered across weeks (i.e., 3 sessions/week in weeks 1-3, 2 sessions/week in weeks 4-6, and 1 session/week in weeks 7-9).
  Arms: Experimental Group 2

SUMMARY:
This study will measure the effects of interactive, whole-body video games on movement behavior in people with chronic low back pain.

DETAILED DESCRIPTION:
A fundamental clinical problem in individuals with chronic low back pain is the significant alteration in movement patterns that restrict lumbar spine motion. This restriction of lumbar motion is particularly evident in patients with kinesiophobia; that is, a fear of movement due to possible injury or reinjury. For chronic back pain patients with kinesiophobia it is critical to develop an effective intervention to increase spine motion while minimizing concerns of pain and harm. Accordingly, we have developed a innovative video games that track whole-body motion and are designed to encourage spinal flexion while reducing concerns of pain and harm among individuals with low back pain. Our games have two distinct advantages. First, within this video game environment, visual feedback can be altered by changing the feedback gain of a given movement (e.g., the magnitude of a given joint movement could appear on screen as either larger or smaller than the actual movement). Thus, gain manipulation will result in progressively larger amounts of lumbar spine flexion during game play. Second, video games are potent distractors that can reduce attention to pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Low back pain that has been ongoing for at least half the days in the last 6 months
* Average pain intensity of greater than 3 over the past week on a 0-10 Numerical Rating Scale
* Disability greater than 4 on Roland and Morris Disability Questionnaire
* Agrees with statement "It is not really safe for a person with my back problem to be physically active" or Tampa Scale of Kinesiophobia score greater than 36
* Has sought care or consultation from a health care provider for back pain
* Meets category 1, 2, or 3 on the Classification System of the Quebec Task Force on Spinal Disorders which reflects low back pain without neurological signs
* Working proficiency in English

Exclusion Criteria:

* Has a personal history of the following neurological disorders: Alzheimers, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinsons, Neuropathy, Stroke, Seizures
* Has a personal history of the following cardiorespiratory disorders: Congestive heart failure, heart attack in past 2 years
* Has a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, Muscular Dystrophy, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis
* History of spine surgery or a hip arthroplasty
* Has active cancer
* Has a chronic disease that may restrict movement or preclude safe participation
* Has used opioids within 30 days prior to study enrollment
* Reports being pregnant, lactating, or that they anticipate becoming pregnant within 2-months
* Reports pending litigation related to CLBP
* Has current drug or alcohol use or dependence that, in the opinion of the PIs, would interfere with adherence to study requirements
* Has significant visual impairment that would prevent virtual reality headset use
* Has significant motion sickness that would prevent virtual reality headset use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S Thomas, P.T., Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] France CR, Thomas JS. Virtual immersive gaming to optimize recovery (VIGOR) in low back pain: A phase II randomized controlled trial. Contemp Clin Trials. 2018 Jun;69:83-91. doi: 10.1016/j.cct.2018.05.001. Epub 2018 May 3. PMID 29730393
- See also: The VIGOR Study — https://movr.vcu.edu/participate/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Experimental Group 2
Started | 74 | 80
Completed | 74 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of subjects enrolled in the two arm of the study
Groups:
- Experimental Group 1: Participants will produce progressively larger lumbar flexion excursions at each game level and across treatment sessions.
  Experimental Group 1: Participants will complete 18 intervention visits over 9 weeks with the number of sessions tapered across weeks (i.e., 3 sessions/week in weeks 1-3, 2 sessions/week in weeks 4-6, and 1 session/week in weeks 7-9).
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1 | Experimental Group 2 | Total
Number analyzed (Participants) | 74 | 80 | 154
Age, Customized [Median (Full Range); unit: years] | 37 [18.1 to 60.9] | 41.1 [19.0 to 60.7] | 39.05 [18.1 to 60.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 24 | 30 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 14 | 12 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 24 | 49
  White | 35 | 35 | 70
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 74 | 80 | 154
Median BMI [Median (Full Range); unit: kg/m^2] | 29.9 [16.3 to 54.9] | 26.7 [19.6 to 58.6] | 28.3 [16.3 to 58.6]
Radiating pain [Count of Participants; unit: Participants]
  yes | 52 | 51 | 103
  no | 22 | 29 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pain Reduction on The Numerical Pain Rating Scale (NPRS)
Description: The Numerical Pain Rating Scale (NPRS) is a pain assessment tool that uses a 11 point scale of 0-10 to help patients rate the intensity of their pain: 0: No pain and 10: The worst pain imaginable. The NPRS is the most commonly used unidimensional pain scale. It can be administered verbally or graphically, and patients are asked to select the number that best reflects their pain intensity over the past 24 hours. The smaller the number (closer to 0), the less pain the subject is enduring, and the larger the number, the more pain they are enduring. Percent change in NPRS rather than raw score change may provide more meaningful information regarding a patient's response to pain treatment.
Time Frame: Baseline measure through the 48-weeks post-treatment measure
Population: Study participants who completed this procedure
Measure: Mean (Standard Deviation); unit: percentage change (NPRS)
Arm/Group | Experimental Group 1 | Experimental Group 2
Number analyzed (Participants) | 72 | 78
percentage change (NPRS) | 30.3 (43.2) | 35.2 (33)

2. Primary Outcome: Change in Disability Using the Roland Morris Disability Questionnaire
Description: Roland Morris Disability Questionnaire: A patient taking the survey agrees or disagrees with these statements (Yes/No). The patient is asked to tick a statement when it applies to him that specific day, this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The items of the questionnaire are assessed on a 0-10 numeric rating scale in which 0 means no disability and 10 is maximum disability. The sum of the seven items equals the total score of the PDI, which ranges from 0 to 70, with higher scores (closer to 70) reflecting higher interference of pain with daily activities and a lower score (closer to 0) has less interference of pain with daily activities.. Test-retest reliability 24-item: intraclass correlation (ICC) ranges from 0.42 - 0.91 T
Time Frame: Baseline measurement through 48-weeks post-treatment measurement change
Population: Subjects that completed this procedure
Measure: Mean (Standard Deviation); unit: score on Roland Morris Disability Questi
Arm/Group | Experimental Group 1 | Experimental Group 2
Number analyzed (Participants) | 71 | 77
score on Roland Morris Disability Questi | 37 (34.6) | 25 (35.2)

ADVERSE EVENTS:
Time Frame: The data was collected at baseline through the end of the study procedures, baseline over 9 weeks.
Arm/Group | Experimental Group 1 | Experimental Group 2
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/80
Other Adverse Events (participants affected / at risk) | 4/74 | 3/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group 1 (N=74) | Experimental Group 2 (N=80)
A transient ischemic attack TIA (General disorders) | 1 (1) | 0 (0) — TIA attack, not related to the study
Shoulder work injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Injured should at work, not study related
Knee Bone Spurs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject developed knee bone spurs, not related to the study
micro-discectomy on L5-L5 and a laminectomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — one subject had a micro-discectomy on L5-L5 and a laminectomy, not related to the study
pulled a muscle in his left hip and lower back while changing a car tire (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — One subject pulled a muscle in his left hip and lower back while changing a car tire, not related to the study
back surgery prior to coming in for V2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — one subject had to have back surgery prior to coming in for V2, not related to the study procedures
minor surgery and it turned out to be a major surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — one subject was scheduled for a minor surgery and it turned out to be a major surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03463824/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03463824/ICF_000.pdf